CLINICAL TRIAL: NCT01819194
Title: Contact Lens Comfort Relative to Meibomian Gland Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: CR-5282
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Results first posted 2014-12-09 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-05

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- senofilcon A (Experimental): Acuvvue Oasys with Hydaclear Plus with 38% water.
  Interventions: Device: senofilcon A

INTERVENTIONS:
Device: senofilcon A

SUMMARY:
This trial aims to establish a correlation between patient reported comfort while using soft contact lenses and meibomian gland dysfunction (MGD).

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be able to read, understand, and sign the statement of informed consent and receive a fully executed copy of the form.
2. The subject be able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be 18 and less than 39 years of age.
4. The subject must be an adapted soft contact lens wearer in both eyes (Defined as having been a full times lens wearer for at least 3 months).
5. Subjects must be current full time daily wearers of Acuvue Oasys lenses (defined as, at least 6 hours per day, 5 days per week).
6. The subject's spherical equivalent distance refraction must be in the range of 0.00 to -6.00D in each eye.
7. The subject must present at visit 1 with a current copy of their spectacle prescription.
8. The subject must have the best corrected visual acuity of 0.18 or better in each eye as assessed by LogMAR chart.
9. The subject must have normal eyes (i.e., no ocular medication, or infections of any type)

Exclusion Criteria:

1. Wear Acuvue Oasys with Hydraclear Plus on an extended wear basis.
2. Wear Acuvue Oasys with Hydraclear Plus for astigmatism.
3. History of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia, active or recent varicella, viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva; mycobacterial infection of the eye; and/or fungal disease of the eye.
4. Use of concomitant ocular medications during the study period. Topical artificial tears or contact lens lubricants are allowed, but no instillation on the day of examinations.
5. Any systemic disease, autoimmune disease, or use of medications, which may interfere with contact lens wear.
6. Subjects using medications influencing tear production such as steroids, immunosuppressive agents and/or anti-cholinergics (e.g. cold and allergy medications, tricyclic antidepressants) for treatment of autoimmune connective tissue disease may not be enrolled in this study if they have not been on a stable dosing regimen for 30 days prior to the Eligibility Visit. Subjects may use birth control medications since there is inconclusive evidence relative to the influence on tear film.
7. Any infectious disease (e.g. Hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV, by self report).
8. Subjects reporting discomfort at screening visit related to fit or care system abnormalities (both determined by the investigator), ocular conditions such as conjunctival infections, iritis.
9. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
10. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
11. Entropion, ectropion, extrusion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosion,aphakia, or moderate or above corneal distortion by keratometry.
12. Any previous, or planned, ocular or intraocular surgery (radial keratotomy, LASIK, ETC.)
13. Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g. past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
14. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
15. Monovision or multi-focal contact lens correction
16. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment
17. History of binocular vision abnormality or strabismus
18. History of serious mental illness
19. History of seizures

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fullerton, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 64 subjects were enrolled in this study. Of the enrolled subjects 2 did not meet the eligibility criteria and 62 were dispensed a study lens. Of the dispensed subjects 60 completed the study and 2 were discontinued.
Groups:
- Overall: Subjects only wore one lens: senofilcon A, 38% water. Subjects, were enrolled and screened per inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Overall
Started | 62
Completed | 60
Not Completed | 2
Not completed — Loss of study articles | 2

BASELINE CHARACTERISTICS:
Population: 64 subjects enrolled with 60 Completing
Groups:
- Dispensed Subjects: All subjects that were dispensed the study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.53 (3.050)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Comfort as Measured by the Contact Lens Users Experience Questionnaire (CLUE)
Description: CLUE is survey that is used to assess subjective comfort of the test article. The higher the score the better on a range of 0 to 120.
Time Frame: Post 3 days of wear
Population: Subjects are those who were enrolled, randomized, and completed the study per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Senofilcon A, 38% Water: Senofilcon A, 38% water
Arm/Group | Senofilcon A, 38% Water
Number analyzed (Participants) | 60
units on a scale | 58.67 (18.430)

2. Primary Outcome: Meibbomian Gland Dysfunction (MGD)as Measured by MGD Scale
Description: Meibomian Gland Dysfunction (MGD) as measured using the MGD 0 - 11 scale translated into grades 0 to 3 where 0 refers to absence of markers.
Time Frame: Post 3 days of wear
Population: Subjects analyzed are those who enrolled, randomized, and completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Senofilcon A, 38% Water
Number analyzed (Participants) | 60
Number analyzed (Eyes) | 120
eyes
  Grade 0 | 0
  Grade 1 | 88
  Grade 2 | 32
  Grade 3 | 0

ADVERSE EVENTS:
Time Frame: Data was collected over the course of the study, approximately 1 week.
Arm/Group | Senofilcon A, 38% Water
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less